CLINICAL TRIAL: NCT01126086
Title: An Open-label Pharmacokinetic, Pharmacodynamic and Tolerability Study of Otamixaban Given as a Single 80 μg/kg Bolus Plus 100 μg/kg/h Continuous Infusion for 24 Hours in Subjects With Mild and Moderate Hepatic Impairment, and in Matched Subjects With Normal Hepatic Function.
Brief Title: Pharmacokinetic, Pharmacodynamic and Tolerability Study of Otamixaban in Patients With Mild and Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP6207; U1111-1116-8891 (Other: UTN)
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild impairment (Experimental): Patients with mild hepatic impairment
  Interventions: Drug: otamixaban XRP0673
- Moderate impairment (Experimental): Patients with moderate impairment
  Interventions: Drug: otamixaban XRP0673
- Healthy subjects (Experimental): Matched healthy subjects
  Interventions: Drug: otamixaban XRP0673

INTERVENTIONS:
Drug: otamixaban XRP0673 — Pharmaceutical form: solution for injection
  Route of administration: intravenous

SUMMARY:
Primary Objective:

- To study effect of mild and moderate hepatic impairment on the pharmacokinetics of otamixaban.

Secondary Objective:

- To assess the pharmacodynamic effects of otamixaban on subjects with mild and moderate hepatic impairment and in matched subjects with normal hepatic function.

DETAILED DESCRIPTION:
The duration of each part of the study for one subject was 28 days of screening, 1 day of treatment, with 5 days in the unit (Day -1 to Day 4) and a 8 to 11 days of follow-up after start of infusion.

ELIGIBILITY:
Inclusion criteria:

- Subjects with hepatic impairment:

* Body weight between 50.0 kg and 115.0 kg inclusive if male, between 40.0 kg and 100.0 kg inclusive if female, Body Mass Index between 18.0 and 34.9 kg/m2 inclusive
* Stable chronic liver disease assessed by medical history, physical examination, laboratory values
* Vital signs, cardiac function and laboratory parameters within the acceptable range for subjects with hepatic impairment
* If female, subject must use a double contraception method, except if she is sterilized for more than 3 months or postmenopausal
* Patients with hepatic impairment will be matched to healthy subjects who are defined as healthy by physical examination, medical history and laboratory findings and are matched to patients with respect to age, gender, and body weight. Inclusion/exclusion criteria for healthy subjects may differ slightly from those listed for patients and are defined in the study protocol

Exclusion criteria:

* Uncontrolled clinically relevant cardiovascular, pulmonary, gastrointestinal, metabolic, hematological, neurological, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness
* Creatinine level above the upper limit of normal
* Hepatocarcinoma
* Acute hepatitis
* Hepatic encephalopathy grade 2, 3 and 4
* History or presence of drug or alcohol abuse within two years before inclusion
* Smoking more than 15 cigarettes or equivalent per day, unable to refrain from smoking during the institutionalization
* Any significant change in chronic treatment medication within 14 days before inclusion

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
PK parameters including Ceoi, AUClast, AUC, C1min, CL, Vss, and t1/2z | Day 1 to Day 4
Pharmacodynamic based on coagulation parameters, activated partial prothrombin time (aPTT), prothrombin time (PT), and international normalized ratio (INR) | Screening (-28 days) up to 4 days after treatment

SECONDARY OUTCOMES:
Safety based on treatment-emergent adverse events, clinical laboratory evaluations, vital signs, and ECG | Screening (-28 days) up 8 to 11 days after treament

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Investigational Site Number 840003, Miami Gardens, Florida
  - Investigational Site Number 840001, Orlando, Florida
  - Investigational Site Number 840002, Knoxville, Tennessee